CLINICAL TRIAL: NCT00670657
Title: CRITIC: Phase II Pilot Multicenter Study on Efficacy and Safety of Liposomal Amphotericin B (AmBisome®) at 2 mg/kg/Day in the Treatment of Candidemia and Invasive Candidiasis in Non-Neutropenic Patients
Brief Title: CRITIC - Treatment of Candidemia and Invasive Candidiasis
Acronym: CRITIC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Luigi Antonio Picaro, Gilead Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GS-IT-131-0177
Record Dates: First submitted 2008-04-29; First posted 2008-05-02 (Estimated); Last update posted 2009-03-27 (Estimated); Status verified 2009-03

CONDITIONS: Candidemia; Invasive Candidiasis
Keywords: candidemia; invasive candidiasis; Ambisome; liposomal amphotericin B
MeSH Terms: conditions — Candidemia; Candidiasis, Invasive | interventions — liposomal amphotericin B

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): AmBisome® 2 mg/kg/day in a unique daily IV administration
  Interventions: Drug: AmBisome

INTERVENTIONS:
Drug: AmBisome — Patients will receive 2mg/kg/day IV daily administration of AmBisome® over 30-60 minutes as a reaction to signs/symptoms and positive Candida culture

SUMMARY:
Patients will receive 2mg/kg/day IV daily administration of AmBisome® over 30-60 minutes as a reaction to signs/symptoms and positive Candida culture

DETAILED DESCRIPTION:
Subjects will be enrolled to receive intravenously AmBisome® at 2 mg/kg/day for a maximum of 4 weeks. Treatment will be discontinued in case of failure, adverse events precluding treatment or success. In case of success AmBisome® at 2 mg/kg/day should be administered for at least 5 days after the complete resolution of all clinical findings of an active infection or for at least 8 days after the last positive blood culture or culture from a normally sterile site. It is not recommended to declare failure (and therefore change treatment) before giving at least 5 days of antifungal therapy. Failures in patients given less than 5 days of treatment should be well documented (e.g. persistent positive cultures despite catheter removal, clinical deterioration in absence of any explanation other than the fungal infection). Follow-up evaluations will be conducted at 2 and 4 weeks after the end of AmBisome® therapy. At end of treatment (time point for success or failure) patients may be shifted to oral (not intravenous) antifungals at the discretion of the local investigator, once a complete response has been achieved, if secondary prophylaxis is deemed necessary.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to ICU for all medical reasons that meet the inclusion criteria
* Males or non pregnant females (women of child-bearing potential must have a negative serum or urine pregnancy test at baseline).
* Subjects who are 14 years old or older.
* Subjects with at least one positive blood culture isolation of a Candida spp. from a specimen or from a normally sterile site (including abdominal catheters), drawn within 96 hours prior to study entry.
* Subjects who have clinical evidence of infection AT SOME TIME WITHIN 48 HOURS PRIOR TO ENROLLMENT, including AT LEAST ONE of the following:

  1. temperature> 38°C on 2 occasions at least 4 hours apart or one determination greater than 38.5°C (internal, at oesophagus, tympani or bladder levels).
  2. systolic blood pressure < 90, or a >30 mm Hg decrease in systolic BP from the subject's normal baseline.
  3. Signs of inflammation (swelling, heat, erythema, purulent drainage) from a site infected with Candida
* Subjects or their legal representative (but the subject should sign it in any case when able to) must sign a written informed consent form. Written informed consent must be obtained before any study-related procedure is carried out.

Exclusion Criteria:

* Subjects with a history of allergy or intolerance to AmBisome®
* Subjects who have received systemic antifungal therapy within 15 days prior to inclusion in the study
* Any severe cardiovascular disease (such as arrhythmias, in particular) which may constitute a contra-indication to AmBisome® administration
* Subjects with an absolute neutrophil count of less than 500/mm3 in the 48 hours before enrolment in the study
* Subjects with a diagnosis of AIDS (positive HIV serology in association with either CD4 cell counts < 200 cells/mm3or history of an opportunistic infection /neoplasm), aplastic anemia, or Chronic Granulomatous Disease.
* Subjects with moderate or severe liver disease defined as any one or more of the following:

  * Alkaline phosphatase, ALT, AST, or total bilirubin greater than 5 times the ULN (upper limit of normal)
* Subjects with a severe renal impairment defined by a serum creatinine of more than 2.5 mg/dL.
* Women who are pregnant or breastfeeding.
* Subjects who are unlikely to survive more than 24 hours.
* Subjects who previously participated in this study.
* Subjects who have received within the two weeks before study entry, are receiving or likely to receive any investigational drug (unlicensed new chemical entity).

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2007-05; Primary Completion 2008-12 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Success at End of Trial (EOT) - Success is defined as: The definition of success is (criteria a, b, c and d must be satisfied): a. i) Absence of all clinical signs and symptoms present at baseline and absence of any new signs and symptoms that may be | Through 4 weeks

SECONDARY OUTCOMES:
Efficacy at the 2nd and 4th week after the end of therapy | Through 4th week
Safety of the 2 mg/kg/day regimen | Through 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Luigi Picaro, Study Director — Gilead Sciences
Locations (1):
- Gilead Sciences Srl, Milan, Italy